CLINICAL TRIAL: NCT03959995
Title: Effects of an Optimized 13-month Physical Exercise on (Early)-Postmenopausal Risk Factors in Women With Osteopenia and Osteoporosis (Actlife)
Brief Title: Effects of Physical Exercise on Postmenopausal Risk Factors in Women With Osteopenia
Acronym: ACTLIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ER_ACTLIFE
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Osteopenia, Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding attempt of participants by sham exercise. Outcome assessors were unaware of participant's group status (exercise or control) and were not allowed to ask correspondingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): Exercise group
  Interventions: Other: High Intensity Resistance (HIT-RT) and Endurance exercise (HIIT)
- control (Sham Comparator): active control group
  Interventions: Other: Wellness

INTERVENTIONS:
Other: High Intensity Resistance (HIT-RT) and Endurance exercise (HIIT) — Ambulatory, consistently supervised group exercise training (3 training sessions of 40-45 min/week each). 10-12-week blocks of non-linearly periodized high intensity resistance and high impact aerobic dance exercises (HIT-setting) intermitted by 4-6-week periods of endurance-type exercise with high volume and lower intensity. Indi-vidualized training schedules for the RT-section.
  Arms: exercise
Other: Wellness — control group: 3x 10 week blocks, 1 training session/week à 45 min; stretching, light functional gymnastics, yoga with less strengthening techniques over 13 months.
  Arms: control

SUMMARY:
Menopause usually have a serious impact on a woman's life, associated with negative consequences for health and quality of life. Early preventive assessments are very difficult to implement due to the complex hormone-deficiency-induced effects on a large variety of organs and systems with estrogen receptors. In fact, only a few types of interventions have the potential to comprehensively improve the various risk factors and complaints of the menopausal transition. In detail, however, not every form of exercise training or every training protocol is effective for exerting positive effects on selected risk factors. In particular, the training concept for addressing musculoskeletal or cardio-metabolic risk factors differ fundamentally.

In several studies, we confirmed the effect of different complex training programs on risk factors of different postmenopausal female cohorts with special consideration of osteoporotic aspects. The training programs applied in this context were characterized by the consistent implementation of recognized training principles and an in general exercise intensity-oriented approach. Recent studies confirmed the effectiveness of this proceeding for women with relevant postmenopausal risk factors including low bone strength. However, the crucial issue of the most effective, feasible and easily customizable training protocol for addressing postmenopausal risk factors remains to be answered, taking into account that the majority of exercise programs were realized in an ambulatory group setting.

The aim of the study will be to evaluate the effects of an optimized physical training on risk factors and complaints of (early) postmenopausal women with special consideration of the osseous fracture risk.

Note (05.06.2020): Of importance, the intervention has to be cancelled due to COVID-19 lockdown in March 2020 after 13 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* (early)postmenopausal women, ( normal menopause, 1-5 years post)
* Osteopenia and osteoporosis at the lumbar spine or femoral neck Bone Mineral Density (BMD) <-1.0 standard deviation (SD) T-Score, WHO)

Exclusion Criteria:

* BMD <-4.0 SD T-Score (BMD threshold for pharmaceutical therapy according to Dachverband Osteologie (DVO) guideline (mandatory for Germany, Austria, Suisse) for woman 50-60 years).
* Prevalent clinical, low-trauma fractures
* Diseases and drugs with relevant effects on bone and muscle metabolism (e.g. glucocorticoids >7.5 mg/d or bisphosphonate therapy); individual case assessment
* Diseases and drugs with relevant effects on cardiometabolic risk factors (e.g. severe hypertension with corresponding medical therapy); individual case assessment
* Severe cardiovascular events (e.g. stroke, coronary infarction) in the past.
* Other conditions, diseases that exclude exercise training in a group (≤10 persons).

Ages: 48 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — early postmenopausal
Enrollment: 27 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
BMD Lumbar Spine | from baseline to 13 month follow-up
  Bone Mineral Density (BMD) at the lumbar spine region of interest as determined by Dual Energy x-Ray Absorptiometry (DXA)

SECONDARY OUTCOMES:
BMD total Hip | from baseline to 13 month follow-up
  Bone Mineral Density at the total hip region of interest as determined by DXA
Para-vertebral muscle density | from baseline to 13 month follow-up
  Muscle density at the para-vertebral region as determined by Magnetic Resonance Imaging (MRI)
Mid-thigh muscle density | from baseline to 13 month follow-up
  Muscle density at the mid-thigh region as determined by MRI
Metabolic Syndrome | from baseline to 13 month follow-up
  Metabolic Syndrome Z-Score according to the Internationale Diabetes Federation (IDF)
Visceral body fat | from baseline to 13 month follow-up
  Visceral body fat as determined by Magnetic Resonance Imaging (MRI)
Total body fat | from baseline to 13 month follow-up
  Total body fat as determined by whole body DXA
Total Lean Body Mass | from baseline to 13 month follow-up
  Total Lean Body Mass as determined by whole body DXA
Menopausal complaints | from baseline to 13 month follow-up
  Menopausal complaints as determined by the Menopause Rating Scale (German version. Questionnaire with 11 items; scale from 0 (no complaints/problems) to 4 (very severe complaints/problem)
Maximum leg strength | from baseline to 13 month follow-up
  Maximum isokinetic leg extensor strength as determined by an isokinetic leg press
Total fat rate | from baseline to 13 month follow-up
  Total fat rate as determined by Bio Impedance technique (BIA)
Fat free mass | from baseline to 13 month follow-up
  Fat free mass as determined by BIA

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hettchen, MSc, Principal Investigator — Institute of Medical Physics, University of Erlangen-Nürnberg, Germany
Locations (1):
- Institute of Medical Physics, Friedrich Alexander University Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jungmann S, Hettchen M, Kohl M, Kemmler W. Impact of 3 months of detraining after high intensity exercise on menopause-related symptoms in early postmenopausal women - results of the randomized controlled actlife project. Front Sports Act Living. 2023 Jan 5;4:1039754. doi: 10.3389/fspor.2022.1039754. eCollection 2022. PMID 36685065